CLINICAL TRIAL: NCT01989559
Title: A Pilot Study to Assess the Immunologic Response to Booster Vaccination With a Modified gp100 Melanoma Peptide (209-2M) Vaccine in Previously Vaccinated HLA-A2.1+ Patients With Melanoma
Brief Title: Booster Vaccination in Preventing Disease Recurrence in Previously Vaccinated Patients With Melanoma That Has Been Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2013-02097; NCI-2013-02097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PPMC-IRB-02-63; NCI-5925; CDR0000258479; 02-63 (Other: Providence Portland Medical Center); 5925 (Other: CTEP); R21CA099265 (NIH); NCT00052988 (obsolete NCT alias)
Record Dates: First submitted 2013-11-18; First posted 2013-11-21 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2013-11

CONDITIONS: Recurrent Melanoma; Stage IA Skin Melanoma; Stage IB Skin Melanoma; Stage IIA Skin Melanoma; Stage IIB Skin Melanoma; Stage IIC Skin Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Protein Subunit Vaccines; Peptides

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine with Montanide ISA 51 VG or Montanide ISA 51 SC on day 1 and between days 25-30. After 6 months, patients free of disease receive booster injections every 6 months for 3 years in the absence of unacceptable toxicity or disease progression.
  Interventions: Biological: gp100:209-217(210M) Peptide Vaccine; Biological: HPV 16 E7:12-20 Peptide Vaccine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: gp100:209-217(210M) Peptide Vaccine — Given SC
Biological: HPV 16 E7:12-20 Peptide Vaccine — Given SC
  Other Names: HPV-16 E7(12-20) peptide; HPV-16E7(12-20) peptide vaccine; HPV16 E7(12-20) peptide; HPV16 E7(12-20) peptide vaccine
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies booster vaccination in preventing disease recurrence in previously vaccinated patients with melanoma that has been removed by surgery. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Giving booster vaccinations may make a stronger immune response and prevent or delay the recurrence of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the toxicity of booster vaccination with the gp100 (gp100:209-217(210M) peptide vaccine) and human papilloma virus (HPV) peptides in Montanide ISA 51 or Montanide ISA 51 VG administered >= 12 months after the last immunization.

II. To measure the T-cell response to the modified gp100: 209-217 (210M) peptide and the unmodified native gp100 peptide following booster vaccination >= 12 months after the last immunization.

III. To measure the T-cell response to the control human leukocyte antigen (HLA)-A2 restricted clusters of differentiation (CD)8 epitope of papilloma virus HPV16E7:12-20 following booster vaccination >= 12 months after the last immunization.

IV. To perform detailed studies of the memory T cells persisting >= 12 months after immunization.

OUTLINE:

Patients receive gp100:209-217(210M) peptide vaccine and HPV 16 E7:12-20 peptide vaccine with Montanide ISA 51 VG or Montanide ISA 51 subcutaneously (SC) on day 1 and between days 25-30. After 6 months, patients free of disease receive booster injections every 6 months for 3 years in the absence of unacceptable toxicity or disease progression.

After completion of study treatment, patients are followed up at 6 months, every 6 months for 5 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed treatment on protocol 99-9 [T98-0081] "A Randomized Phase II Trial to Determine the Immune Response to a Mutated gp100 Melanoma Peptide Vaccine in HLA-A2.1+ Patients with a > 1mm Melanoma on Initial Biopsy;" patients are not required to have received every planned vaccine as long as the reason for stopping was not disease progression or dose limiting toxicity
* Patients must be >= 12 months from their last vaccination with gp100 and be free of melanoma; patients who have remained continuously free of disease and patients who have had a recurrence that has been completely resected (stage IV no evidence of disease [NED]) are eligible
* Patients must have a good performance status (Karnofsky performance status [PS] 80-100)
* White blood cells (WBC) >= 3500/mm^3
* Platelets (plt) >= 100,000/mm^3
* Hemoglobin >= 9 gm/100 ml
* Serum creatinine =< 2 mg/dl
* Total bilirubin =< 2.0 mg/dl
* Patients must have recovered from any effects of major surgery and be free of significant systemic infection
* Women of childbearing potential must have a negative pregnancy test and must avoid becoming pregnant while on treatment; men must avoid fathering a child while on treatment
* Patients must give written informed consent prior to initiation of therapy
* Patients with a history of psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy

Exclusion Criteria:

* Patients must not have clinically detectable melanoma
* Patients who require or are likely to require systemic corticosteroids for intercurrent illness are ineligible
* Patients with any significant medical disease other than the melanoma, which in the opinion of the investigator would significantly increase the risk of immunotherapy, are ineligible
* Patients should be free of any other cancers or deemed at low risk for their recurrence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percentage of positive CD8+ T cells | Up to 11 years
  Characterized using three different in vitro assays. Fresh and cryopreserved peripheral blood mononuclear cells (PBMC) will be analyzed for gp100 peptide-specific CD8+ T cells using a fluorescinated, modified gp100, peptide-specific, A2-restricted tetramer binding assay and the interferon (IFN) gamma specific enzyme-linked immunosorbent spot (ELISPOT) and cytokine flow cytometry (CFC) assays.
Change in CD8+ T cell frequency | Up to 11 years
  Differences in immune parameters will be graphically depicted by means of density plots, frequency histograms, box and whisker-plots, dot-plots, trellis graphics (where appropriate) and other plots and graphs. Analyses of continuous variables will be performed first on the original frequency data. Goodness of fit statistics will be employed to determine whether assumptions underlying test statistics (e.g., normality) are satisfied. If assumptions for the test procedures are violated, then rank-transformed or arcsin-transformed data will be used. Probability tests will be two-sided.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Urba, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States